CLINICAL TRIAL: NCT03439917
Title: Effect of Carnitine Supplementation on Liver Steatosis, Insulin Sensitivity, Plasma Glucose Homeostasis, Skeletal Muscle Metabolism and Energetics: a Pilot Study
Brief Title: Effects of Carnitine Supplementation on Liver and Muscle
Acronym: ECLIPSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 17086; 17/EM/0441 (Other: REC Reference)
Record Dates: First submitted 2018-02-14; First posted 2018-02-20 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Insulin Resistance
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Insulin Resistance | interventions — slif protein, Drosophila; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carnitine and Meal Replacement Drink (Experimental): 2g L-carnitine tartrate consumed with a meal replacement milkshake (Slimfast, UK) twice a day for 24 weeks.
  Interventions: Dietary Supplement: L-Carnitine tartrate; Dietary Supplement: Meal Replacement Drink
- Placebo and Meal Replacement Drink (Placebo Comparator): 2g Maltodextrin consumed with a meal replacement milkshake (Slimfast, UK) twice a day for 24 weeks.
  Interventions: Dietary Supplement: Meal Replacement Drink; Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: L-Carnitine tartrate — 2g L-Carnitine tartrate as a powder consumed twice a day
  Arms: Carnitine and Meal Replacement Drink
Dietary Supplement: Meal Replacement Drink — 325ml dairy-based meal replacement drink ('Slimfast' trademark of KSF Acquisition UK Ltd) consumed twice a day
  Other Names: Slimfast
Dietary Supplement: Maltodextrin — 2g Maltodextrin powder packaged to mimic carnitine powder consumed twice a day
  Arms: Placebo and Meal Replacement Drink

SUMMARY:
It will be evaluated whether carnitine, a dietary supplement, reduces liver fat and improves metabolism in individuals who have a high concentration of fat within their liver. Participants will be given either Carnitine or placebo, together with a meal replacement milkshake twice daily for 6 months.

DETAILED DESCRIPTION:
NAFLD occurs when too much fat accumulates in liver tissue. This can, over time, cause inflammation and scarring of the liver, eventually leading to chronic liver disease and cirrhosis. It is strongly associated with diabetes and obesity, both of which are endemic in Western societies.

Carnitine enables cells in the body to use fat as a fuel, and recent studies have suggested that carnitine supplementation may reduce liver triglyceride content. Muscle and liver are the major sites in the body which coordinate glucose and fat metabolism. As well as assessing the effect of carnitine supplementation on liver fat, its effect on metabolic processes within these tissues will also be measured

ELIGIBILITY:
Inclusion Criteria:

* Elevated liver fat on screening abdominal ultrasound
* Capable of providing informed consent
* Non-vegetarian diet
* BMI <40 kg/m2
* Weekly ethanol consumption <21 units/week
* Negative non-invasive liver screen, including Hepatitis B and C serology, liver autoantibodies, transferrin saturation, α1-antitrypsin levels.

Exclusion Criteria:

* Known history of cardiovascular disease
* Known diabetes mellitus
* Known psychiatric comorbidity
* Chronic kidney disease
* Surgery within 6 months prior to start of study
* Exposure to drugs known to influence hepatic steatosis (including steroids, statins, omega-3-fatty acids)
* Current smokers
* Contraindications to magnetic resonance scanning, including implanted ferrous material (implantable pacemakers or defibrillators), metallic ocular foreign bodies, ferromagnetic aneurysm clips or severe claustrophobia.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Intrahepatic triglyceride (IHTG) content | 24 weeks
  IHTG measured by proton magnetic resonance spectroscopy

SECONDARY OUTCOMES:
liver sensitivity to insulin | 24 weeks
  suppression of glucose output from the liver during a 20 mU.m-2.min-1 hyperinsulinaemic euglycaemic clamp
whole body insulin sensitivity | 24 weeks
  whole body glucose uptake during a 50 mU.m-2.min-1 hyperinsulinaemic euglycaemic clamp
Muscle lipid content | 24 weeks
  lipid content of the vastus lateralis muscle measured by proton magnetic resonance spectroscopy
Skeletal muscle sensitivity to insulin | 24 weeks
  Arterialised-venous vs. femoral venous difference in blood glucose concentration during the last hour of a 2 hour 50 mU.m-2.min-1 hyperinsulinaemic euglycaemic clamp
whole body composition | 24 weeks
  Fat and lean tissue mass assessment by dual energy X-ray absorptiometry
Liver energy metabolism | 24 weeks
  hepatic ATP flux assessed by 31-phosphorous magnetic resonance spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Guru Aithal, MD, PhD, Principal Investigator — University of Nottingham
Locations (1):
- David Greenfield Human Physiology Unit, Nottingham, Notts, United Kingdom

IPD SHARING:
Plan to Share IPD: No